CLINICAL TRIAL: NCT05674682
Title: Seroincidence Study Among Men Who Have Sex With Men and Transgender Women - The ImPrEP Seroincidence Study. A Sub-study of Implementation of HIV Pre-exposure Prophylaxis (PrEP) for Men Who Have Sex With Men and Transgender People: A Demonstration Project in the Context of Combined Prevention in Brazil, Mexico and Peru - the ImPrEP Study
Brief Title: Seroincidence Study Among Men Who Have Sex With Men and Transgender Women - The ImPrEP Seroincidence Study
Acronym: Seroincidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evandro Chagas National Institute of Infectious Disease (Other)
Collaborators: Valdiléa Veloso dos Santos, Ph.D. (Unknown); Beatriz Grinzstejn, MD, PhD (Unknown); Brenda Hoagland, MD, PhD (Unknown); Celia Landmann Szwarcwald, PhD (Unknown); Thiago Torres, PhD (Unknown); Maria Cristina Pimenta, MD, PhD (Unknown); Marcos Benedetti, MA (Unknown); Marília Santini Oliveira (Unknown); Ronaldo Ismério Moreira, PhD (Unknown); Sandro Nazer Coutinho (Unknown); Sylvia Lopes Maia Teixeira, PhD (Unknown); Nilo Martínez Fernandes, PhD (Unknown); Hamid Vega-Ramírez, MD, MSc (Unknown); Sérgio Bautista-Arredondo, MD, PhD (Unknown); René Leyva-Flores, PhD (Unknown); Helleen Vermandere (Unknown); Santiago Ávila-Ríos, PhD (Unknown); Claudia García-Morales, PhD (Unknown); Carlos Cáceres, MD, MPH, PhD (Unknown); Kelika A. Konda, PhD (Unknown); Juan Vicente Guanira, MD, PhD (Unknown); Giovanni Ravasi, MD, MScPH (Unknown)
Responsible Party: Principal Investigator, Raquel Malaguthi de Souza, Regulatory Affairs Associate, Evandro Chagas National Institute of Infectious Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20012619.9.1001.5262
Record Dates: First submitted 2023-01-03; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections; Risk Reduction; Risk Behavior; Risky Health Behavior; STD; HIV Seropositivity; HIV Infection Primary
Keywords: MSM; TGW; Imprep; HIV
MeSH Terms: conditions — HIV Infections; Risk Reduction Behavior; Risk-Taking; Health Risk Behaviors; HIV Seropositivity | interventions — HIV Testing

STUDY DESIGN:
Intervention Model Description: MSM and TGW, aged 18 yo or more
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venipuncture or digital puncture for HIV test (Other): MSM and transgender women aged 18 years or older, willing and able to sign informed consent to accept venipuncture or digital puncture for HIV testing
  Interventions: Procedure: HIV testing

INTERVENTIONS:
Procedure: HIV testing — venipuncture or digital puncture for HIV testing

SUMMARY:
PrEP (pre-exposure prophylaxis) is an effective prevention strategy in which HIV-negative individuals take antiretroviral drugs (tenofovir disoproxil fumarate and emtricitabine - TDF/FTC) to reduce HIV acquisition. Clinical studies have shown that the TDF/FTC combination protects MSM and transgender women against HIV infection. According to the PROUD study, PrEP can decrease the risk of HIV infection among MSM by 86% (90% CI 64-96). The international community recognizes that PrEP can be an additional tool in the framework of a combination prevention package for those most at risk of contracting HIV. Data on HIV incidence among MSM and trans women are largely unknown. In Brazil, Mexico and Peru, data on the incidence of HIV among MSM and trans women are very scarce, limited to small cross-sectional studies.Current methods used to determine HIV-1 incidence have many limitations. These methods include mathematical modeling, retrospective calculations of AIDS case reports, age-based prevalence determinations, and prevalence determinations with multiple rounds of longitudinal surveys to estimate HIV incidence, which require numerous assumptions and inputs and can pose additional challenges in the era of expansion of antiretroviral therapy (ART) and increased survival of HIV-1 infected individuals. On the other hand, prospective longitudinal cohort studies of high-risk individuals can be used to estimate incidence; however, they are often labor-intensive, complex, very expensive, difficult to implement in most countries, and have recruitment biases. Laboratory methods can be unbiased and do not require complicated assumptions and case-by-case weighting. The cross-sectional use of Recent HIV Infection Tests (TRIs) based on biomarkers offers, in principle, accessible, reliable and low risk of bias options for estimating incidence.

ELIGIBILITY:
Inclusion Criteria:

* MSM and transgender women
* aged 18 years or older
* willingness and ability to sign an informed consent form.

Exclusion Criteria:

* Individuals currently using PrEP, PEP or receiving antiretroviral therapy;
* Individuals unable to understand the study or who do not agree to sign the consent form;
* Individuals who are participating in a clinical trial of antiretroviral medication or any investigational product to prevent the acquisition of HIV infection (for example, monoclonal antibodies such as PEP or PrEP)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men having Sex with other Men and Trans Gender Women
Enrollment: 4000 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Identification of recent infections in a given high-risk population (MSM and TGW), including those in defined geographic areas for evaluate epidemics, calibrate models, design and evaluate interventions. | 2 years
  Blood collected for viral load from those with confirmed HIV infection will be used to distinguish recent HIV-1 infections of long-term infections

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Instituto Nacional de Infectologia Evandro Chagas (Fiocruz), Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional de Infectologia Evandro Chagas/ FIOCRUZ, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torres TS, Teixeira SLM, Hoagland B, Konda KA, Derrico M, Moreira RI, Guanira JV, Benedetti M, Nazer S, Calvo GM, Vargas S, Benites C, Bigolin A, Alonso Neto JB, Farias A, Guimaraes Lacerda MV, Raenck Silva DA, Paz LC, Madruga JV, Salvatierra Flores HJ, Boluarte GP, Osco Tamayo CV, Castro Antezana HT, Pimenta MC, Borquez A, Luz PM, Grinsztejn B, Szwarcwald CL, Caceres CF, Veloso VG; ImPrEP Seroincidence Study Group. Recent HIV infection and annualized HIV incidence rates among sexual and gender minorities in Brazil and Peru (ImPrEP seroincidence study): a cross-sectional, multicenter study. Lancet Reg Health Am. 2023 Dec 2;28:100642. doi: 10.1016/j.lana.2023.100642. eCollection 2023 Dec. PMID 38076411
- See also: Baral S, Sifakis F, Cleghorn F, Beyrer C. Elevated risk for HIV infection among men who have sex with men in low- and middle-income countries 2000-2006: a systematic review — http://databank.worldbank.org/data/download
- See also: Beyrer C, Baral SD, van Griensven F, Goodreau SM, Chariyalertsak S, Wirtz AL, et al. Series HIV in men who have sex with men 1 Global epidemiology of HIV infection in men who have sex with men. Lancet — http://dx.doi.org/10.1016/S0140-6736(12)60821-6
- See also: Core Team, 2013. R: A language and environment for statistical computing [Internet]. Vienna: R Foundation for Statistical Computing; 2013. — http://www.r-project.org
- See also: Gomez GB, Borquez A, Caceres CF, Segura ER, Grant RM, Garnett GP, et al. The potential impact of pre-exposure prophylaxis for HIV prevention among men who have sex with men and transwomen in Lima, Peru: a mathematical modelling study. Salomon JA, editor. — http://dx.plos.org/10.1371/journal.pmed.1001323
- See also: Grinsztejn B, Jalil EM, Monteiro L, Velasque L, Moreira RI, Garcia ACF, et al. Unveiling of HIV dynamics among transgender women — http://www.ncbi.nlm.nih.gov/pubmed/2818803
- See also: Silva-Santisteban A, Eng S, de la Iglesia G, Falistocco C, Mazin R. HIV prevention among transgender women in Latin America: implementation, gaps and challenges. J Int AIDS Soc [Internet]. 2016 [cited 2018 Mar 14];19(3 Suppl 2):20799. — http://www.ncbi.nlm.nih.gov/pubmed/27431470
- See also: UNAIDS. Miles to go - closing gaps. Global AIDS update 2018. — https://www.unaids.org/sites/default/files/media_asset/miles-to-go_en.pdf